CLINICAL TRIAL: NCT00853645
Title: Initial Chronic Human Validation Study: Subcutaneous Implantable Cardioverter Defibrillator (S-ICD) System
Acronym: Chronic II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: DN-11398
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Ventricular Tachyarrhythmias
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subcutaneous implantable cardioverter defibrillator (S-ICD) System (Experimental): Single-arm with 6 patients implanted with an S-ICD System
  Interventions: Device: Subcutaneous Implantable Defibrillator (S-ICD) System

INTERVENTIONS:
Device: Subcutaneous Implantable Defibrillator (S-ICD) System

SUMMARY:
Primary objective is to evaluate the safety and performance of the implanted Subcutaneous implantable cardioverter defibrillator (S-ICD) system. A maximum of 10 subjects were to be enrolled and followed for one month to collect data on the safety, efficacy, and performance of the implanted S-ICD system. Additionally, patient comfort will be assessed as will cosmetic outcome.

ELIGIBILITY:
Inclusion Criteria:

* replacement of an existing transvenous implantable cardioverter defibrillator (ICD) system
* American College of Cardiology/American Heart Association/Heart Rhythm Society (ACC/AHA/HRS) Class I or II indications for ICD implantation
* Age >= 18 years
* Appropriate pre-operative Electrocardiogram (ECG) as measured with a specially developed template

Exclusion Criteria:

* Subjects unable or unwilling to provide informed consent
* Any condition which precludes the subject's ability to comply with the study requirements
* Females who are pregnant or lactating and pre-menopausal women who are unwilling to use adequate birth control for the duration of the study
* Participation in another investigational device trial at any time during the conduct of the S-ICD system trial without written consent from the sponsor.
* Patients with a serious medical condition and life expectancy of less than one year.
* Patients with documented spontaneous and frequently recurring ventricular tachyarrhythmias (VT) that is reliably terminated with anti-tachycardia pacing
* Patients with existing epicardial patches or subcutaneous electrodes in the left thoracic quadrant
* Patients with chronic renal failure, i.e. with a creatinine level of >2.5 mg/dl unless prescribed drug therapy known to increase creatinine levels in which case the value should be <= 3mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen O'Connor, PhD, Hon FRACP, Study Director — Boston Scientific Corporation
Locations (2):
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch

REFERENCES:
- [Derived] Bardy GH, Smith WM, Hood MA, Crozier IG, Melton IC, Jordaens L, Theuns D, Park RE, Wright DJ, Connelly DT, Fynn SP, Murgatroyd FD, Sperzel J, Neuzner J, Spitzer SG, Ardashev AV, Oduro A, Boersma L, Maass AH, Van Gelder IC, Wilde AA, van Dessel PF, Knops RE, Barr CS, Lupo P, Cappato R, Grace AA. An entirely subcutaneous implantable cardioverter-defibrillator. N Engl J Med. 2010 Jul 1;363(1):36-44. doi: 10.1056/NEJMoa0909545. Epub 2010 May 12. PMID 20463331

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subcutaneous Implantable Cardioverter Defibrillator (S-ICD) System
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subcutaneous Implantable Cardioverter Defibrillator (S-ICD) System
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.24 (11.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Successful Induced Ventricular Fibrillation Conversion
Description: Sustained ventricular fibrillation induced by the investigator is successfully converted. A successful conversion was defined as two consecutive successful shocks out of four attempts with either standard polarity or with reverse polarity.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Implantable Cardioverter Defibrillator (S-ICD) System
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Subcutaneous Implantable Cardioverter Defibrillator (S-ICD) System: Single-arm with 6 patients implanted with an Subcutaneous implantable cardioverter defibrillator (S-ICD) System
Arm/Group | Subcutaneous Implantable Cardioverter Defibrillator (S-ICD) System
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subcutaneous Implantable Cardioverter Defibrillator (S-ICD) System (N=6)
Severe acute coronary syndrome. (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subcutaneous Implantable Cardioverter Defibrillator (S-ICD) System (N=6)
Pulse generator rotation (Product Issues) | 3 (3)
Inappropriate paced beats post shock (Product Issues) | 1 (1)
Electrode removed and retunneled at implant (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No